CLINICAL TRIAL: NCT02878967
Title: Standardized Long Term Follow-up of Patients After Endovascular Embolization of a Brain
Brief Title: Standardized Long Term Follow-up of Patients After Endovascular Embolization of a Brain Aneurysm
Acronym: ANENDOVASC
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: RBC_2015_14
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Aneurysm
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
The time-frame and the follow-up elements after embolization of brain aneurysm are not standardized. Therefore, few reliable follow-up data are available for these patients.

This study aims at collecting standardized long term data for these patients, in order to assess the occurence of aneurysm recanalization and particularly those requiring another intervention on the aneurysm.

DETAILED DESCRIPTION:
An intracranial aneurysm is a localised dilatation in the wall of an intracranial artery, creating a zone of fragility where the main risk is rupture (meningeal haemorrhage). Intracranial aneurysms are the 1st vascular pathology treated in the NRI department at the Rothschild Foundation (FOR). Since 2002, between 150 and 250 patients have been treated each year using the embolisation technique (filling the aneurysm sac with coils). Over the last thirteen years, this represents the largest cohort in France, with more than 2,000 patients selectively treated for one or more intracranial aneurysms, i.e. more than 2,500 aneurysms. Treatment consists of excluding the aneurysmal cavity from the bloodstream, usually by "plugging" it with platinum metal coils.

After treatment by embolisation of the aneurysm, recanalisation (recirculation of blood in the aneurysm, exposing the patient to a new risk of haemorrhage due to aneurysmal rupture) of the cavity may occur after a few months or years (approximately in 7% of cases). In addition, new aneurysms may develop during the patient's lifetime, often several years later.

Another type of aneurysm treatment is also possible: surgical treatment, which consists of clipping the neck of the aneurysm. Whichever type of treatment is used, patients are monitored according to a protocol for the first year following treatment, with visits at 6 months and 1 year: an MRI is performed 6 months after embolisation. An arteriogram was performed at one year, and a consultation was held for clinical evaluation. A retrospective assessment of follow-up data (study of 2009-2013 files) showed that the date of this consultation varied considerably and that the schedule of follow-up visits over the first 10 years was not standardised, which means that reliable follow-up data are not available for these patients. The occurrence of recanalisation led us to propose standardised longer-term follow-up, with imaging (MRI and/or arteriography) 3 years after the operation. In our clinical experience, this follow-up schedule (at 3-6 months, 1 year and then 3 years) makes it possible to detect recanalisation requiring re-treatment. The aim of this research is to obtain standardised, longer-term follow-up data for a large series of patients who have undergone embolisation or surgical treatment of an intracranial aneurysm.

ELIGIBILITY:
Inclusion Criteria:

* curative embolization of a brain aneurysm
* age >18 years old

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing curative embolization of a brain aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-11-25 (Actual); Primary Completion 2030-11-24 (Estimated); Study Completion 2040-11-24 (Estimated)

PRIMARY OUTCOMES:
long term evaluation of aneurysm occlusion | 5 years after embolization
  Roy classification

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël Blanc, MD, Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France